CLINICAL TRIAL: NCT04800484
Title: The Effects of AFO Heel Height and Stiffness on Gait
Acronym: AFOHeel
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Iowa (Other)
Responsible Party: Principal Investigator, Jason Wilken, Associate Professor, University of Iowa
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 201811701
Record Dates: First submitted 2021-03-11; First posted 2021-03-16 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Musculoskeletal Injury; Musculoskeletal Diseases; Peripheral Nervous System Diseases
Keywords: Gait Analysis; Ankle Foot Orthosis; Biomechanics
MeSH Terms: conditions — Musculoskeletal Diseases; Peripheral Nervous System Diseases

STUDY DESIGN:
Intervention Model Description: Participants will be evaluated in their clinically configured AFO and without an AFO if able. They will also complete evaluation with four provided heel wedge conditions in randomized order: tall soft, tall firm, short soft, short firm.
Who Masked: Participant
Masking Description: Participants will be blinded to the heel wedge conditions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (24):
- Arm 1: (Experimental): Testing Order: Clinical AFO, Tall Soft, Tall Firm, Short Soft, Short Firm, NoAFO
  Interventions: Device: Tall Soft; Device: Tall Firm; Device: Short Soft; Device: Short Firm
- Arm 2: (Experimental): Testing Order: Clinical AFO, Tall Soft, Tall Firm, Short Firm, Short Soft, NoAFO
  Interventions: Device: Tall Soft; Device: Tall Firm; Device: Short Soft; Device: Short Firm
- Arm 3: (Experimental): Testing Order: Clinical AFO, Tall Soft, Short Soft, Tall Firm, Short Firm, NoAFO
  Interventions: Device: Tall Soft; Device: Tall Firm; Device: Short Soft; Device: Short Firm
- Arm 4: (Experimental): Testing Order: Clinical AFO, Tall Soft, Short Soft, Short Firm, Tall Firm, NoAFO
  Interventions: Device: Tall Soft; Device: Tall Firm; Device: Short Soft; Device: Short Firm
- Arm 5: (Experimental): Testing Order: Clinical AFO, Tall Soft, Short Firm, Tall Firm, Short Soft, NoAFO
  Interventions: Device: Tall Soft; Device: Tall Firm; Device: Short Soft; Device: Short Firm
- Arm 6: (Experimental): Testing Order: Clinical AFO, Tall Soft, Short Firm, Short Soft, Tall Firm, NoAFO
  Interventions: Device: Tall Soft; Device: Tall Firm; Device: Short Soft; Device: Short Firm
- Arm 7: (Experimental): Testing Order: Clinical AFO, Tall Firm, Tall Soft, Short Soft, Short Firm, NoAFO
  Interventions: Device: Tall Soft; Device: Tall Firm; Device: Short Soft; Device: Short Firm
- Arm 8: (Experimental): Testing Order: Clinical AFO, Tall Firm, Tall Soft, Short Firm, Short Soft, NoAFO
  Interventions: Device: Tall Soft; Device: Tall Firm; Device: Short Soft; Device: Short Firm
- Arm 9: (Experimental): Testing Order: Clinical AFO, Tall Firm, Short Soft, Tall Soft, Short Firm, NoAFO
  Interventions: Device: Tall Soft; Device: Tall Firm; Device: Short Soft; Device: Short Firm
- Arm 10: (Experimental): Testing Order: Clinical AFO, Tall Firm, Short Soft, Short Firm, Tall Soft, NoAFO
  Interventions: Device: Tall Soft; Device: Tall Firm; Device: Short Soft; Device: Short Firm
- Arm 11: (Experimental): Testing Order: Clinical AFO, Tall Firm, Short Firm, Tall Soft, Short Soft, NoAFO
  Interventions: Device: Tall Soft; Device: Tall Firm; Device: Short Soft; Device: Short Firm
- Arm 12: (Experimental): Testing Order: Clinical AFO, Tall Firm, Short Firm, Short Soft, Tall Soft, NoAFO
  Interventions: Device: Tall Soft; Device: Tall Firm; Device: Short Soft; Device: Short Firm
- Arm 13: (Experimental): Testing Order: Clinical AFO, Short Soft, Tall Soft, Short Firm, Tall Firm, NoAFO
  Interventions: Device: Tall Soft; Device: Tall Firm; Device: Short Soft; Device: Short Firm
- Arm 14: (Experimental): Testing Order: Clinical AFO, Short Soft, Tall Soft, Tall Firm, Short Firm, NoAFO
  Interventions: Device: Tall Soft; Device: Tall Firm; Device: Short Soft; Device: Short Firm
- Arm 15: (Experimental): Testing Order: Clinical AFO, Short Soft, Tall Firm, Short Firm, Tall Soft, NoAFO
  Interventions: Device: Tall Soft; Device: Tall Firm; Device: Short Soft; Device: Short Firm
- Arm 16: (Experimental): Testing Order: Clinical AFO, Short Soft, Tall Firm, Tall Soft, Short Firm, NoAFO
  Interventions: Device: Tall Soft; Device: Tall Firm; Device: Short Soft; Device: Short Firm
- Arm 17: (Experimental): Testing Order: Clinical AFO, Short Soft, Short Firm, Tall Soft, Tall Firm, NoAFO
  Interventions: Device: Tall Soft; Device: Tall Firm; Device: Short Soft; Device: Short Firm
- Arm 18: (Experimental): Testing Order: Clinical AFO, Short Soft, Short Firm, Tall Firm, Tall Soft, NoAFO
  Interventions: Device: Tall Soft; Device: Tall Firm; Device: Short Soft; Device: Short Firm
- Arm 19: (Experimental): Testing Order: Clinical AFO, Short Firm, Tall Soft, Tall Firm, Short Soft, NoAFO
  Interventions: Device: Tall Soft; Device: Tall Firm; Device: Short Soft; Device: Short Firm
- Arm 20: (Experimental): Testing Order: Clinical AFO, Short Firm, Tall Soft, Short Soft, Tall Firm, NoAFO
  Interventions: Device: Tall Soft; Device: Tall Firm; Device: Short Soft; Device: Short Firm
- Arm 21: (Experimental): Testing Order: Clinical AFO, Short Firm, Tall Firm, Short Soft, Tall Soft, NoAFO
  Interventions: Device: Tall Soft; Device: Tall Firm; Device: Short Soft; Device: Short Firm
- Arm 22: (Experimental): Testing Order: Clinical AFO, Short Firm, Tall Firm, Tall Soft, Short Soft, NoAFO
  Interventions: Device: Tall Soft; Device: Tall Firm; Device: Short Soft; Device: Short Firm
- Arm 23: (Experimental): Testing Order: Clinical AFO, Short Firm, Short Soft, Tall Firm, Tall Soft, NoAFO
  Interventions: Device: Tall Soft; Device: Tall Firm; Device: Short Soft; Device: Short Firm
- Arm 24: (Experimental): Testing Order: Clinical AFO, Short Firm, Short Soft, Tall Soft, Tall Firm, NoAFO
  Interventions: Device: Tall Soft; Device: Tall Firm; Device: Short Soft; Device: Short Firm

INTERVENTIONS:
Device: Tall Soft — Tall heel wedge made of soft foam
  Other Names: TS
Device: Tall Firm — Tall heel wedge made of firm foam
  Other Names: TF
Device: Short Soft — Short heel wedge made of soft foam
  Other Names: SS
Device: Short Firm — Short heel wedge made of firm foam
  Other Names: SF

SUMMARY:
The proposed study evaluates the effect of ankle foot orthosis (AFO) heel height and stiffness on the forces and motion of the lower limb during over-ground walking in individuals who use an AFO for daily walking. Previous studies suggest that heel height and stiffness effect limb loading, but these data and the analysis techniques applied are limited. In this study, heel cushions with different height and stiffness's (4 conditions) will be placed in participants shoes and they will walk at controlled and self-selected speeds. Participants will also walk with their AFO as configured prior to enrollment, and with no AFO if possible. The proposed study will provide evidence that can be used by clinicians and researchers to align braces that most effectively improve function during every-day walking.

DETAILED DESCRIPTION:
In this study the investigators to evaluate the effect of ankle foot orthosis (AFO) heel height and stiffness on the forces and motion of the lower limb during over-ground walking in individuals who use an AFO for daily walking. Previous studies suggest that heel height and stiffness effect limb loading, but these data and the analysis techniques applied are limited.

Two groups of subjects with impairments below the knee, that result in functional deficits and require daily AFO use, will be recruited for this study. The first group will have unilateral deficits associated with musculoskeletal injury or disease (Group 1), and the second group will have bilateral or unilateral deficits associated with peripheral nervous system disease (Group 2).

Lower limb forces and body motion will be assessed using computerized motion capture and force plates in the floor, as individuals walk over-ground. Small reflective markers placed on the participant's skin and force measuring plates in the floor will be used. Participants will walk with their clinically provided AFO, with added heel cushions of two different heights and stiffness's (4 conditions) at a controlled velocity and self-selected velocity. If able, they will walk without their AFO at a self-selected pace. Participants will be asked to provide information regarding their health condition and opinions of the conditions tested.

ELIGIBILITY:
GROUP 1 Patient Inclusion criteria

* Ages: 18-70
* Daily AFO use to address unilateral, below knee functional deficits that result from limb injury or musculoskeletal disease (e.g. fracture, muscle and/or nerve injury, ankle arthritis)
* Greater than 2 weeks using their current AFO
* Ability to walk 50 feet without use of an assistive device (Cane, crutch, etc.)
* Ability to walk at a slow to moderate pace
* AFO fits into traditional footwear
* Able to read and write in English and provide written informed consent

GROUP 1 Patient Exclusion criteria

* Pain > 6/10 while walking during testing or an increase in pain during testing of > 2/10.
* Central Nervous System disorder or disease (e.g. Stroke, Cerebral Palsy, Spinal Cord Injury, or other conditions that result in lower limb spasticity).
* Disorder or disease that affects peripheral nerve function (e.g. diabetes, Charcot Marie Tooth).
* Limited contralateral lower limb function due to injury or neurological/musculoskeletal disorder.
* Use of a hinged/articulating AFO (e.g. Plantar flexion stop, Dorsiflexion assist/stop, free motion), Charcot Restraint Orthotic Walker (CROW) boot, AFOs that restrict all motion in the ankle and foot.
* Use of an AFO that crosses the knee (Knee brace)
* Insufficient space in shoe to accommodate the tallest heel wedge and their AFO
* Visual or hearing impairments that limit walking ability or could limit the ability to comply with instructions given during testing
* Pregnancy - Per participant self-report. Due the expected small number of pregnant individuals, and resulting inability to account for its effect on resulting outcomes participants will be withdrawn from the study.
* Body Mass index > 40.

GROUP 2 Patient Inclusion Criteria

* Ages: 18-70
* Daily AFO use to address below knee functional deficits that result from disease involving the peripheral nervous system (e.g. Charcot Marie Tooth, Multiple Sclerosis, diabetes)
* Greater than 2 weeks using their current AFO (unilateral or bilateral)
* Ability to walk 50 feet without use of an assistive device (Cane, crutch, etc.)
* AFO fits into traditional footwear
* Ability to walk at a slow to moderate pace
* Able to read and write in English and provide written informed consent

GROUP 2 Patient Exclusion Criteria

* Pain > 6/10 while walking or an increase in pain during testing of > 2/10
* Central Nervous System disorder or disease (e.g. Stroke, Cerebral Palsy, Spinal Cord Injury, or other conditions that result in lower limb spasticity)
* Limited function due to limb injury (e.g. fracture, muscle and/or nerve injury)
* Use of a hinged/articulating AFO (e.g. Plantar flexion stop, Dorsiflexion assist/stop, free motion), Charcot Restraint Orthotic Walker (CROW) boot, AFOs that restrict all motion in the ankle and foot.
* Use of an AFO that crosses the knee (Knee brace)
* Insufficient space in shoe to accommodate the tallest heel wedge and their AFO
* Visual or hearing impairment that limit walking ability or limit the ability to comply with instructions given during testing
* Pregnancy - Per participant self-report. Due the expected small number of pregnant individuals, and resulting inability to account for its effect on resulting outcomes participants will be withdrawn from the study
* Body Mass index > 40.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-11-07 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Center of pressure velocity timing | Baseline
  Timing of peak center of pressure velocity (percent stance) during gait.
Center of pressure velocity magnitude | Baseline
  Magnitude of peak center of pressure velocity (m/s) during gait.
Modified Socket Comfort Score (Comfort) | Baseline
  Comfort scores range from 0 = most uncomfortable to 10 = most comfortable.
Modified Socket Comfort Score (Smoothness) | Baseline
  Smoothness scores range from 0 = least smooth to 10 = most smooth.
Numerical Pain Rating Scale | Baseline
  Pain will be assessed using a standard 11-point numerical pain rating scale, in which 0 = no pain and 10 = worst pain imaginable.
Participant wedge preference | Baseline
  The participant will rank order their preference for their Clinical AFO, Tall Soft, Tall Firm, Short Soft, or Short Firm wedge on a questionnaire.

SECONDARY OUTCOMES:
Ankle Range of Motion | Baseline
  Ankle range of motion (degrees) during gait.
Peak Ankle Moment | Baseline
  Peak ankle moment (Nm/kg) during gait.
Peak Ankle Power | Baseline
  Peak ankle power (W/kg) during gait.

OTHER OUTCOMES:
Activities-Specific Balance Confidence (ABC) | Baseline
  The ABC provides a standardized evaluation of balance confidence across a range of common daily tasks.
PROMIS Patient reported outcomes for physical function | Baseline
  The Patient Reported Outcome Information System (PROMIS) physical function Computer Adaptive Test (CAT) is a computerized assessment measuring physical function. It is scored using a T-score in which 50 is the mean of a relevant reference population and 10 is the standard deviation (SD) of that population. In a given PROMIS domain, a T-score above 50 represents more of the measured variable than the population average.

CONTACTS AND LOCATIONS:
Overall Officials: Jason M Wilken, PT, PhD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No